CLINICAL TRIAL: NCT06822036
Title: PROSPECTIVE RANDOMIZED CONTROLLED TRIAL EVALUATING the EFFICACY of INTRAOPERATIVE ARISTA™ AH POLYSACCHARIDE APPLICATION on the POSTOPERATIVE BLOOD LOSS in PATIENTS UNDERGOING ROBOTIC ASSISTED RADICAL PROSTATECTOMY for the TREATMENT of PROSTATE CANCER
Brief Title: EFFICACY of INTRAOPERATIVE ARISTA POLYSACCHARIDE APPLICATION on the POSTOPERATIVE BLOOD LOSS in PATIENTS UNDERGOING RARP for the TREATMENT of PROSTATE CANCER
Acronym: ARISTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital Gronau (Other)
Collaborators: Becton, Dickinson and Company (Industry); University of Leipzig (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-601-f-S
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer (Adenocarcinoma); Blood Loss, Postoperative; Erectile Function
Keywords: prostate cancer; blood loss; potency rates; ARISTA™ AH
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma; Postoperative Hemorrhage; Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm B - no periooperative application of 5g of ARISTA™ AH (No Intervention): No perioperative application of ARISTA™ AH to the prostate bed and neurovascular bundles at the end of the surgery; no other hemostyptic agent in aforementioned area; (ARISTA™ AH application outside of aforementioned areas are allowed; e.g. to the fossa obturatoria)
- Arm A - periooperative application of 5g of ARISTA™ AH (Active Comparator): Perioperative application of 5g of ARISTA™ AH to the prostate bed and neurovascular bundles during and at the end of the surgery to control bleeding and oozing in accordance with labelled directions; no other hemostyptic agent in aforementioned area
  Interventions: Procedure: Arm A - Application of 5g of ARISTA™ AH

INTERVENTIONS:
Procedure: Arm A - Application of 5g of ARISTA™ AH — Perioperative application of 5g of ARISTA™ AH to the prostate bed and neurovascular bundles during and at the end of the surgery to control bleeding and oozing in accordance with labelled directions; no other hemostyptic agent in aforementioned area
  Arms: Arm A - periooperative application of 5g of ARISTA™ AH

SUMMARY:
Background and aim of the study: Radical prostatectomy (RP) is one of the most commonly used treatment options for localized prostate cancer (PCa). Blood loss and deterioration of erectile function is, however, a common unwanted side effect of RP. Previous series demonstrated that the robot-assisted RP (RARP) approach is associated with lower blood-loss rates than open RP. However, several factors might contribute to higher blood loss rates at RARP: First, ileus still represents a major complication. To further reduce complication rates of postoperative ileus most high-volume centers lower the intraabdominal pressure during RARP, which in turn might lead to higher estimated blood loss rates. Second, to improve functional outcomes such as erectile function and early recovery of urinary continence, many surgeons perform intrafascial nerve sparing, which is considered a dissection that follows the periprostatic fasica and allows a whole-thickness preservation of the neurovascular bundles. Ideally, many surgeons aim to avoid thermal application in favor of optimal nerve sparing quality. Moreover, partial or complete secondary resection in context of intraoperative frozen section protocols such as NeuroSafe might further increase risk of blood loss. Taken together, to enable best balance between low intraabdominal pressure as primary prevention of postoperative ileus, maximum nerve sparing quality (i.e. intrafascial approach) and low blood loss rates, atraumatic and athermal hemostatic measures such as polysaccharide application are needed. Thus, we perform a multicenter randomized controlled prospective study with superiority trial design, in which such hemostat agent is applied to the neurovascular bundle areas. We examine if such agent leads to a relevant clinical improvement indicated by higher postoperative hemoglobin levels compared to the control group. As an exploratory co-primary endpoint of interest, we examine erectile function after RARP. Erectile dysfunction (ED) after RP is caused by several different mechanisms and commonly multifactorial. However, one of the main reasons for ED after RP is injury to the cavernous nerves during surgery. Currently, nerve-sparing surgical approaches are commonly performed, if oncologically appropriate, to minimize postoperative potency decline. Notwithstanding improvements of nerve-sparing techniques, a certain degree of nerve damage during surgery is inevitable. In order to keep the rates of postoperative ED at a minimum, it is reasonable to stabilize the cavernous nerves during surgery. In a previous pilot conducted by Chedid et al, the polysaccharide ARISTA™ AH was applicated on the cavernous nerves during robot-assisted RP (RARP) to optimize hemostasis. Later analysis of the study results revealed unexpectedly high potency rates in those men. This observation raised the question, if ARISTA™ AH may have the potential to stabilize the cavernous nerves and thus ameliorate postoperative potency rates. As the previous study by Chedid et al was originally not designed for this endpoint and did not have a control group, we are planning to evaluate this question as a meaningful exploratory co-primary endpoint in the same study cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age range ≥ 45 to ≥68 yrs
* Biopsy proven prostate cancer treated with robotic-assisted radical prostatectomy
* Intrafascial nerve sparing surgery (unilaterally or bilaterally)
* Preoperative urinary continence
* Group A Preoperative unassisted International Index of Erectile function (IIEF)-5 score range 8-16 (i.e. moderate (8-11) and mild to moderate (12-16))

Exclusion Criteria:

* Severe intellectual limitations preventing to fully understand the study concept and its content
* High risk prostate cancer (PSA ≥ 20 ng/ml or biopsy Gleason-Score ≥ 8 or suspected T4)
* Suspected bone or visceral metastases at preoperative imaging Neoadjuvant androgen deprivation therapy
* Any prior local therapy of the prostate (including subvesical deobstruction or radiation therapy)
* Any prior chemotherapy or colon/rectal surgery
* Any prior pelvic trauma that required surgical intervention
* Depression or other psychological or neurological disease (dementia, schizophrenia, bipolar disorder etc.)
* Peyronie's disease
* Polyneuropathia
* IPSS Score >19 and QoL >3
* Bilateral secondary (complete or partial) resection of the neurovascular bundle
* No contraindications for phosphodiesterase type 5 inhibitor intake (i.e. suited for most penile rehabilitation regimes)
* Any endocrine function disorder (not including diabetes)

SURGICAL AND PERIOPERATIVE EXLUSION CRITERIA:

* Accessory pudendal arteries (APA) preservation, if an APA is identified
* For a) nerve sparing and b) controlling bleeding in the area of the prostate bed and neurovascular bundles after prostate removal, no monopolar thermal application are allowed but suturing and clip application is allowed. For secondary resection of the neurovascular bundle and controlling bleeding, mono- or bipolar thermal application, clip application and suturing is allowed.
* No surgical revision within 7d after RARP (Clavien Dindo classified complication ≥3b)
* No definitive anastomotic partial or complete rupture (identified via cystogram within 30d after RARP)

Ages: 45 Years to 68 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 362 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
postoperative blood loss | improvement in ΔHgB between day 5-6 day and preoperative hemoglobin levels
  In theory, the experimental treatment should not have any improvement in ΔHgB between day 5-6 day and preoperative hemoglobin levels
comparison between groups A and B concerning the unassisted IIEF-5 score between groups | 3, 6 and 12 months after RARP
  A difference of the median IIEF-5 score of minimally four points between groups is considered as clinically relevant. Based on these considerations, 84 patients per treatment arm are required (including an assumed dropout rate of 33% or less). As it is possible that the effect of nerve stabilization of ARISTA™ AH may differ according to the preoperative potency status, two groups of patients will be analyzed:

CONTACTS AND LOCATIONS:
Overall Officials: Sami-Ramzi Leyh-Bannurah, PD, Principal Investigator — Klinik für Urologie, Urologische Onkologie und Roboter-assistierte Chirurgie
Locations (3):
- Germany (3):
  - Martini Klinik am UKE GmbH, Hamburg, Hamburg
  - St. Antonius-Hospital Gronau GmbH, Klinik für Urologie, Urologische Onkologie und Roboter-assistierte Chirurgie, Gronau, North Rhine-Westphalia
  - Klinik und Poliklinik für Urologie des Universitätsklinikums Leipzig, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: No